CLINICAL TRIAL: NCT06498492
Title: Early Versus Delayed Laparoscopic Cholecystectomy For Acute Mild Biliary Pancreatitis: A Prospective Comparative Study
Status: Completed | Type: Observational
Sponsor: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Responsible Party: Principal Investigator, Ishwor Thapaliya, Mr., Tribhuvan University Teaching Hospital, Institute Of Medicine.
Other Study IDs: 180(6-11)E2
Record Dates: First submitted 2024-07-05; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Biliary Acute Pancreatitis
Keywords: Biliary Acute Pancreatitis; Laparoscopic Cholecystectomy; Outcomes
MeSH Terms: interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early cholecystectomy group: For group division patients were asked to select a paper randomly from a box, offering them the choice between early or delayed laparoscopic cholecystectomy although the ultimate decision was influenced by patient preference. Those patients whose paper came early underwent early laparoscopic cholecystectomy within index hospital.
  Interventions: Procedure: Laparoscopic Cholecystectomy
- Late cholecystectomy group: Those patients whose paper came delayed were discharged after symptoms subside and were readmitted after 6 weeks to undergo laparoscopic cholecystectomy.
  Interventions: Procedure: Laparoscopic Cholecystectomy

INTERVENTIONS:
Procedure: Laparoscopic Cholecystectomy — Laparoscopic cholecystectomy (LC) has been established as the gold standard of treatment for acute mild biliary pancreatitis.

SUMMARY:
The goal of this observational study is to evaluate the outcomes of early versus delayed cholecystectomy following mild biliary pancreatitis in Nepalese patients.

DETAILED DESCRIPTION:
This was a hospital-based prospective observational study performed at a tertiary academic center from September 2020 to August 2021.

Patients diagnosed with acute mild biliary pancreatitis according to the Revised Atlanta classification 2012 were enrolled from the Emergency/Outpatient Department. Detailed history taking and thorough general and systemic examinations were conducted. Eligible patients were informed about treatment options (early vs. delayed LC) and provided informed written consent. Randomization into "early" or "delayed" groups was performed, and detailed investigations were conducted. To avoid bias, randomization was accomplished by lottery method. In the early group, laparoscopic cholecystectomy was performed during the same admission, while delayed group patients underwent surgery after symptom resolution and readmission. Surgeries were performed under general anesthesia with standard laparoscopic techniques with surgeons of equivalent qualifications. Postoperative care included analgesics and antibiotics, with follow-up examinations and histopathological assessments conducted at specified intervals. Oral intake and pain management protocols were implemented postoperatively, with patients monitored for recovery and instructed to return to normal activities after staple removal. Patients were asked to complete a visual analog pain score (VAS) from 0 (no pain) to 10 (intolerable pain) on the seventh postoperative day.

ELIGIBILITY:
Inclusion Criteria:

* Patients (>18 years of age) who presented with the diagnosis of acute mild biliary pancreatitis in our hospital were included after obtaining written consent

Exclusion Criteria:

* patients with severe sepsis, acute moderate and severe pancreatitis, immunocompromised conditions, biliary peritonitis, cholangitis, pregnancy, admission to the intensive care unit (ICU) or high dependency unit (HDU) and those who declined to provide consent.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with acute mild biliary pancreatitis according to the Revised Atlanta classification 2012 were enrolled from the Emergency/Outpatient Department.Eligible patients were informed about treatment options (early vs. delayed LC) and provided informed written consent. Randomization into "early" or "delayed" groups was performed, and detailed investigations were conducted. To avoid bias, randomization was accomplished by lottery method. In the early group, laparoscopic cholecystectomy was performed during the same admission, while delayed group patients underwent surgery after symptom resolution and readmission.
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-02-12 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
Total duration of hospital stay among early cholecystectomy group vs delayed cholecystectomy group | 4 weeks
  In the early group, the time interval between admission to the day of discharge following laparoscopic cholecystectomy was taken into account. In the delayed group, total duration of hospital stay in conservative management period as well as for laparoscopic cholecystectomy was taken into account.

CONTACTS AND LOCATIONS:
Locations (1):
- Ishwor Thapaliya, Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: Yes
Types of IPD to be Shared:
  Demographic data of the participants (age, gender, comorbidities). Data on the severity of biliary pancreatitis. Surgical outcomes, including the length of hospital stay, duration of surgery, and conversion rate to open cholecystectomy.
  Data on recurrent biliary events and perioperative complications.
  Groups and Time Frame:
  The study divided participants into two groups:
  Early Cholecystectomy Group:
  Intervention: Underwent laparoscopic cholecystectomy within a short period after diagnosis of acute mild biliary pancreatitis.
  Time Frame: Mean hospital stay of 5.42 ± 1.01 days.
  Delayed Cholecystectomy Group:
  Intervention: Underwent laparoscopic cholecystectomy after an extended period following the initial diagnosis.
  Time Frame: Mean hospital stay of 9.36 ± 1.53 days.
  Data Sharing Mechanism:
  Data will be available upon reasonable request from the corresponding author.
Supporting Information: Study Protocol
Time Frame: Data will be available for a period of 1 year.
Access Criteria: Researchers must provide a clear scientific rationale for requesting the data. Data will be shared upon reasonable request to the corresponding author. Requests must detail the intended use of the data and ensure it aligns with the ethical guidelines, ensuring patient confidentiality.